CLINICAL TRIAL: NCT03498482
Title: Treating Posttraumatic Stress Disorder and Reducing Aggressive Behavior in Street Children and Vulnerable Children in Burundi Using Narrative Exposure Therapy for Forensic Offender Rehabilitation.
Brief Title: Adressing PTSD Symptoms and Aggressive Behavior in Vulnerable Children in Burundi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry); Psychologues sans Frontières Burundi (Other); Université Lumière de Bujumbura (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal investigator, University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKCR17
Record Dates: First submitted 2017-12-22; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Posttraumatic Stress Disorder; Aggressive Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FORNET (Experimental): During FORNET, the client, with the assistance of the therapist, constructs a chronological narrative of his or her entire life with a focus on exposure to traumatic stress and committed violence. Empathic understanding, active listening, congruency and unconditional positive regard are key components of the therapist's behavior. The therapist asks in detail for the client's emotions, cognitions, physiological reactions, and sensory informations during traumatic and aggressive events to link them to an autobiographical context, namely time and place. In total the individuals receive 8 sessions of FORNET, every session lasting between 1.5 and 2 hours depending on the needs of the participant.
  Interventions: Behavioral: Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET)

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET) — FORNET aims to reduce trauma-related symptoms and aggressive behavior via narrative exposure of traumatic and violent life events.

SUMMARY:
Children either living in the streets of Bujumbara or that are similarly affected by extreme poverty or violence are regularly exposed to traumatic events. Additionally, they often find themselves in situations where engaging in violent behavior appears to be useful or even necessary for survival. The Narrative Exposure Therapy for violent offenders (FORNET) aims to reduce both PTSD symptoms and aggressive behavior. It helps the children to anchor fearful experiences and potential positive emotions linked to violent behaviour in the past. Additionally, visions for the future are developed in order to enable reintegration into the family.

The investigators want to provide evidence, that FORNET effectively reduces PTSD symptoms and ongoing aggressive behavior which in change facilitates reintegration into society.

ELIGIBILITY:
Inclusion Criteria:

* High degree of symptoms of posttraumatic stress disorder according to UCLA PTSD Reaction Index

Exclusion Criteria:

* Psychotic symptoms

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change of load of traumatic symptoms measured via the UCLA Adolescent PTSD Index (PTSD scale administered by Clinicians) | baseline; 5 months follow-up; 9 months follow-up

SECONDARY OUTCOMES:
Change of number of aggressive acts measured via an adaption of the Domestic and Community Violence Checklist | baseline; 5 months follow-up; 9 months follow-up
Change of experienced shame measured via the Shame Variability Questionnaire | baseline; 5 months follow-up; 9 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- vivo international & Psychologues sans Frontières mental health center, Bujumbura, Bujumbura Mairie Province, Burundi

IPD SHARING:
Plan to Share IPD: No